CLINICAL TRIAL: NCT03263286
Title: Home Therapy for Upper Limb Stroke Rehabilitation Using the HandSOME Exoskeleton
Brief Title: Home Therapy for Stroke Rehabilitation Using the HandSOME Exoskeleton
Acronym: HandSOME
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: The Catholic University of America (Other)
Collaborators: MedStar National Rehabilitation Network (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016-064
Record Dates: First submitted 2017-08-21; First posted 2017-08-28 (Actual); Last update posted 2020-08-28 (Actual); Status verified 2020-08

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- HandSOME (Experimental): The intervention is given to this group.
  Interventions: Device: HandSOME

INTERVENTIONS:
Device: HandSOME — Participants use the HandSOME orthosis daily for 8 weeks.

SUMMARY:
This research will evaluate the potential for a novel hand orthosis (HandSOME) to help stroke victims regain functional use of their hand and regain independent living. Participants will use the HandSOME at home regularly for 8 weeks. Clinical evaluations will measure changes from the intervention after the 8 weeks and also at a 3 month followup.

DETAILED DESCRIPTION:
After stroke, individuals often have great difficulty with using the affected hand in functional tasks. The hand frequently suffers from finger flexor hypertonia as well as finger extensor weakness. This leads to increased difficulty in grasp and release of objects. HandSOME is a light weight wearable hand orthosis that increases range of motion and decreases effort during grasping tasks. The goal of this study is to evaluate the HandSOME device's effectiveness in the rehabilitation of stroke patients through an 8 week intervention. Eligible subjects will use the device daily at home for 8 weeks with one visit per week to the clinic to evaluate progress and troubleshoot problems with the device. The hypotheses are that the gains from the 8 weeks of training will be statistically significant and clinically important (defined as gains of greater than 10% of full scale) in the domains of impairment, function and amount of arm use.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of stroke more than six months prior to entry into the study
2. Impaired ability to open affected the hand
3. At least trace ability to extend the wrist and fingers

Exclusion Criteria:

1. Have cognitive deficits that could negatively affect their ability to complete the protocols as evidenced by a score of 24 or less on the Folstein Mini-Mental State Examination
2. Have excessive pain in any joint of the affected extremity that could limit ability to cooperate with the protocols
3. Have serious uncontrolled medical problems as judged by the project therapist
4. Receiving oral or injected antispasticity medications during study treatment
5. MCP and IP passive extension limit > 30 degrees from full extension
6. Excessive tone in the fingers and thumb as determined by Ashworth scores >=3

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2017-04-15 (Actual); Primary Completion 2019-10-07 (Actual); Study Completion 2019-10-07 (Actual)

PRIMARY OUTCOMES:
Change in Fugl-Meyer Test of Arm Function | Change from baseline Fugl-Meyer score at 2 months
  clinical test of arm motor ability and impairment
Change in Action Research Arm Test | Change from baseline Action Research Arm Test score at 2 months
  clinical test of the functional limitations of the upper extremities
Change in Motor Activity Log | Change from baseline Motor Activity Log score at 2 months
  assess the amount and quality of limb use at home

SECONDARY OUTCOMES:
Change in Fugl-Meyer Test of Arm Function at followup | Change from baseline Fugl-Meyer score at 5 months
  clinical test of arm motor ability and impairment
Change in Action Research Arm Test at followup | Change from baseline Action Research Arm Test score at 5 months
  clinical test of the functional limitations of the upper extremities
Change in Motor Activity Log at followup | Change from baseline Motor Activity Log score at 5 months
  assess the amount and quality of limb use at home

CONTACTS AND LOCATIONS:
Locations (1):
- MedStar National Rehabilitation Network, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tianyao Chen, Lum PS. Hand rehabilitation after stroke using a wearable, high DOF, spring powered exoskeleton. Annu Int Conf IEEE Eng Med Biol Soc. 2016 Aug;2016:578-581. doi: 10.1109/EMBC.2016.7590768. PMID 28324934